CLINICAL TRIAL: NCT02593929
Title: Pharmacodynamic Effects and Predictive Biomarkers of JAK/STAT Inhibition With Ruxolitinib in Operable Head and Neck Cancer: a Window Trial
Brief Title: Pharmacodynamic Effects and Predictive Biomarkers With Ruxolitinib in Operable Head and Neck Cancer
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCI 14-207
Record Dates: First submitted 2015-10-14; First posted 2015-11-02 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: squamous cell carcinoma; head and neck cancer; operable
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell; Head and Neck Neoplasms | interventions — ruxolitinib

ARMS (1):
- ruxolitinib (Experimental): Ruxolitinib will be taken orally for 14-21 days prior to surgery, every morning and every evening, and will be discontinued after the morning dose on the day of planned surgical resection.
  Interventions: Drug: ruxolitinib

INTERVENTIONS:
Drug: ruxolitinib

SUMMARY:
This study will identify baseline and/or pharmacodynamic biomarkers of response to ruxolitinib, based upon association with quantitative change in tumor size following 14-21 days of neoadjuvant ruxolitinib in patients with operable HNSCC.

DETAILED DESCRIPTION:
In this study, ruxolitinib will be administered for a short period of 2-3 weeks prior to planned surgical resection of HNSCC. The dose will be 20 mg twice daily, the FDA-approved dose in myelofibrosis. The brief treatment duration is within the expected window of time that elapses from initial patient evaluation by a surgeon to performance of surgery. In the phase 0 or window trial model, a paired specimen analysis permits ex vivo evaluation of target modulation and pharmacodynamic changes in downstream or parallel molecular pathways.32 This study design is optimal in order to assess the biochemical and immunomodulatory effects of ruxolitinib on HNSCC. Furthermore, predictive biomarkers can be developed as related to a clinical endpoint or a biochemical, pharmacodynamic endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed, primary or recurrent, head and neck squamous cell carcinoma, including variants. Patients must have at least one measureable lesion in accordance with RECIST 1.1 (tumor diameter ≥ 1 cm; short-axis lymph node diameter ≥ 1.5 cm) OR by caliper measurement (tumor diameter ≥ 1 cm). Any diagnostic pretreatment biopsy sample is acceptable including FNA.
2. Primary tumors of any head and neck (oral cavity, oropharynx, hypopharynx, or larynx) site will be included.
3. Surgical resection of head and neck must be planned, either as primary treatment or salvage. Patients must undergo research biopsy prior to receiving drug.
4. Age ≥ 18 years.
5. ECOG performance status 0-2 (See Appendix I).
6. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test (sensitivity ≤ 25IU HCG/L) within 4 weeks prior to registration and will be repeated within 72 hours prior to the start of study drug administration.
7. Persons of reproductive potential must agree to use and utilize an adequate method of contraception throughout treatment and for at least 12 weeks after study drug is stopped. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
8. Adequate hematologic, renal and hepatic function, as defined by:

   1. Absolute neutrophil count (ANC) ≥ 1,500/ul, platelets ≥ 150,000/ul.
   2. Creatinine ≤ 1.5 x institutional upper limit of normal (ULN).
   3. Bilirubin ≤ 1.5 x ULN, AST or ALT ≤ 2.5 x ULN.
9. Have signed written informed consent

Exclusion Criteria:

1. Subjects who fail to meet the above criteria.
2. Prior therapy for head and neck cancer is allowed, and the number of treatments is not limited. However, any systemic therapy should have been completed at least 30 days prior to study enrollment. Any radiation to the head and neck should have been completed at least 30 days prior to study enrollment. Palliative radiation outside of the head and neck does not require a washout.
3. Pregnancy or breastfeeding. Women (patients or partners of male patients) of childbearing potential (WOCBP) must practice acceptable methods of birth control to prevent pregnancy. All WOCBP MUST have a negative pregnancy test within 4 weeks prior to registration, and this must be repeated within 72 hours prior to first receiving ruxolitinib. If the pregnancy test is positive, the patient must not receive ruxolitinib and must not be enrolled in the study.
4. Any unresolved chronic toxicity ≥ grade 2 from previous anticancer therapy (except alopecia and anemia), according to Common Terminology Criteria for Adverse Events v4.0 (CTCAE).
5. Current active infection requiring systemic antibiotic or antifungal therapy.
6. Acute hepatitis or known HIV.
7. Treatment with a non-approved or investigational drug within 30 days prior to Day 1 of study treatment.
8. New York Heart Association (NYHA) Class III or IV heart disease.
9. History of thromboembolic event or other condition currently requiring anticoagulation with warfarin (coumadin). Patients who are treated with low molecular weight heparin or fondaparinux are eligible.
10. History of significant bleeding disorder unrelated to cancer, including: diagnosed congenital bleeding disorders (e.g., von Willebrand's disease, diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies, or ongoing or recent (≤ 3 months) significant gastrointestinal bleeding
11. Concomitant Medications, any of the following should be considered for exclusion: Strong CYP3A4 inhibitors: (Patients must discontinue drug 7 days prior to starting ruxolitinib), including but not limited to boceprevir, clarithromycin, conivaptam, indinavir, itraconazle, ketoconazole, lopinavir, mibefradil, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, or voriconazole. In addition, patients will be instructed to avoid grapefruit or grapefruit juice, starfruit, or seville oranges.
12. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
baseline and/or pharmacodynamic biomarkers of response to ruxolitinib based upon association with change in tumor size | 14-21 days

SECONDARY OUTCOMES:
preliminary efficacy of neoadjuvant ruxolitinib in patients with operable HNSCC as determined by quantitative ΔTumor size | 14-21 days
the tolerability of brief neoadjuvant exposure to ruxolitinib as determined by the number of participants with treatment related adverse events as assessed by CTCAE v4.0 | 14-21 days
the effect of ruxolitinib on the tumoral Ki-67 proliferation index | 14-21 days
  Evaluate the change in the KI-67 proliferation index after exposure to ruxolitinib. Ki-67 immunohistochemistry will be performed with the Dako North America M7240 antibody and scored quantitatively with Aperio computer-assisted digital analysis by the research pathologist. In keeping with international consensus guidelines, at least 5000 tumor cells/specimen will be counted. The percentage of positive tumor cells represents the proliferation index.
additional candidate biomarkers of ruxolitinib response or resistance in HNSCC patients as determined by quantitative ΔTumor size | 14-21 days